CLINICAL TRIAL: NCT00036257
Title: Dose-Escalating and Safety Study of CP-461 in Patients With Chronic Lymphocytic Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Collaborators: Cell Pathways (Industry); OSI Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Masking: None | Purpose: Treatment
Other Study IDs: OSI-461-010
Record Dates: First submitted 2002-05-08; First posted 2002-05-09 (Estimated); Last update posted 2011-10-17 (Estimated); Status verified 2011-10

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: Chronic Lymphocytic Leukemia; Leukemia; CLL
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia | interventions — (5-fluoro-2-methyl-1-(4-pyridyl)methylene-3-(N-benzyl)-indene)-acetamide hydrochloride

INTERVENTIONS:
Drug: CP-461

SUMMARY:
The purposes of this study are to determine a maximum tolerated dose and to evaluate the safety and efficacy of CP-461 in patients with Chronic Lymphocytic Leukemia.

ELIGIBILITY:
Inclusion Criteria:

1. Relapsed or refractory chronic lymphocytic leukemia.
2. Patients must have either intermediate or high risk chronic lymphocytic leukemia according to the Rai Staging System.
3. Must have failed at least 1 prior chemotherapy regimen (at least 1 of which included fludarabine) for CLL.
4. No prior therapy within 4 weeks prior to entering the study. Patients must have fully recovered from the acute effects of prior therapy.
5. Platelet count = 75,000/mm3 , hemoglobin = 8 gm/dL.
6. Expected remaining life span > or = three months.
7. ECOG performance status 0 - 2.
8. 18 years or of legal age.
9. Male patients or non-pregnant and non-lactating female patients, who are either using adequate birth control, are surgically sterile or post-menopausal.
10. Negative serum pregnancy test, if fertile female.
11. Willingness and ability to sign an informed consent document.

Exclusion Criteria:

1. Evidence of CNS involvement.
2. Other active malignancy or history of treatment of any malignancy (excluding non-melanoma skin cancer) within the previous three years.
3. Previous therapy with Campath.
4. Patients with low-risk chronic lymphocytic leukemia according to the Rai Staging System.
5. Concurrent immunotherapy.
6. Concurrent use of steroids.
7. Use of an investigational medication or device within 1 month of initiating study therapy.
8. Patients who have had allogeneic bone marrow transplantation.
9. Total serum bilirubin above the upper limit of normal; serum creatinine above the upper limit of normal.
10. AST or ALT > 2.5 times the upper limit of normal.
11. Any condition or any medication which may interfere with the conduct of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15
Dates: Start 2002-03; Study Completion 2003-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Cancer Centers of Florida, Orlando, Florida
  - Albany Regional Cancer Center, Albany, New York
  - Mary Crowley Medical Research Center (US Oncology), Dallas, Texas
  - Tyler Cancer Center, Tyler, Texas
  - Cancer Care Northwest, Spokane, Washington